CLINICAL TRIAL: NCT05128591
Title: An Open-label, Randomized, Single-dose, 2-sequence, 2-period, Crossover, Phase 1 Study Under Fed State to Evaluate the Safety and Pharmacokinetics of AD-109 in Healthy Male Volunteers
Brief Title: A Study to Compare Pharmacokinetic Parameters and Safety Profiles Between AD-109 and AD-1091
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Addpharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AD-109BE
Record Dates: First submitted 2021-11-10; First posted 2021-11-22 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2021-11

CONDITIONS: Embolism and Thrombosis
MeSH Terms: conditions — Embolism and Thrombosis | interventions — Rivaroxaban; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A-Rivaroxaban (Experimental): Period 1 : Reference Drug(AD-1091) Period 2 : Test Drug(AD-109)
  Interventions: Drug: Rivaroxaban 18mg Oral Tablet; Drug: Rivaroxaban 20 MG Oral Tablet
- Arm B-Rivaroxaban (Experimental): Period 1 : Test Drug(AD-109) Period 2 : Reference Drug(AD-1091
  Interventions: Drug: Rivaroxaban 18mg Oral Tablet; Drug: Rivaroxaban 20 MG Oral Tablet

INTERVENTIONS:
Drug: Rivaroxaban 18mg Oral Tablet — AD-109 (Rivaroxaban 18mg) Oral Tablet
Drug: Rivaroxaban 20 MG Oral Tablet — AD-1091 (Rivaroxaban 20mg) Oral Tablet

SUMMARY:
Primary endpoint of this study is to evaluate the pharmacokinetic characteristics of AD-109 in healthy male subjects.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety profiles of AD-109 compared with AD-1091 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body weight equal to or greater than 50kg and Body mass index (BMI) between 18.0 kg/m2 and 30.0 kg/m2 at the time of screening visit
* The Age equal to or greater than 19 in healthy male volunteers at the time of screening visit

Exclusion Criteria:

* Patients with Medical history increasing the risk of bleeding

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2021-11-09 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | pre-dose to 34 hours
  Cmax of Rivaroxaban
Area Under the Curve in time plot (AUCt) | pre-dose to 34 hours
  AUCt of Rivaroxaban

CONTACTS AND LOCATIONS:
Locations (1):
- H+ Yangji Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No